CLINICAL TRIAL: NCT02770768
Title: Flibanserin and Women With Hypoactive Sexual Desire Disorder: A Double-Blind, Randomized, Electrical Neuroimaging Study
Brief Title: Effects of Flibanserin on the Pre- and Post-menopausal Female Brain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution cannot be contacted.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB16-0087
Record Dates: First submitted 2016-04-22; First posted 2016-05-12 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: HSDD (Hypoactive Sexual Desire Disorder); EEG (Electroencephalogram)
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flibanserin (Active Comparator): Drug: Flibanserin
  * 8 weeks
  * 100mg once daily at bedtime
  Interventions: Drug: Flibanserin
- Placebo (Placebo Comparator): Drug: Matching Placebo Matching placebo capsules taken in same amount of pills as the active medication (for 8 weeks once daily at bedtime)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flibanserin — Observational study using electroencephalogram (EEG) and eye movement tracking device at baseline, week 4, and week 8 while subjects are taking either Flibanserin or matching placebo.
  Other Names: Addyi
  Arms: Flibanserin
Drug: Placebo — Observational study using electroencephalogram (EEG) and eye movement tracking device at baseline, week 4, and week 8 while subjects are taking either Flibanserin or matching placebo.
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of the present study is to understand the neurobiological mechanisms of action underlying sexual desire building on prior work Dr. Stephanie Cacioppo has done in which desire was not manipulated. In the present project, Dr. Stephanie Cacioppo is manipulating desire through Flibanserin (Addyi) vs. placebo and she will be measuring subjective sexual desire as a manipulation check. The investigators will address this goal using a double-blind randomized outpatient design and determine the pre-post neurobehavioral change in the Flibanserin group and investigate the extent to which Flibanserin normalizes brain activity in premenopausal women with HSDD and the extent to which regional brain activation is associated with changes in symptoms and behavior (as measured with self-report measures of sexual desire and/or eye-tracking movements).

DETAILED DESCRIPTION:
Hypoactive sexual desire disorder (HSDD) is the most common sexual complaint in women. Over the past 8 years, Dr. Stephanie Cacioppo has developed and validated the Desire Intention task, in which individuals are instructed to indicate as rapidly and as accurately as possible whether or not each visually presented stimulus (e.g., attractive persons of the opposite sex) is sexually desirable to them at the moment of the experiment. Flibanserin (Addyi) is a new medication approved by the FDA for the treatment of HSDD in pre-menopausal women. The investigators propose a study using the DIT to determine the extent to which Flibanserin normalizes brain activity in women with HSDD and the extent to which regional brain activation is associated with changes in symptoms and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 21-45 or 51-74
* Pre- or Postmenopausal
* DSM-5 diagnosis of hypoactive sexual desire disorder (HSDD)
* Right-handed

Exclusion Criteria:

* Male
* Pregnant women
* Nursing women
* Post-menopausal women
* Women who report not being able to stop drinking alcohol during the duration of the study
* Currently taking psychotropic medication
* History of seizures or neurological disorders
* Under hormonal therapy
* Current or past diagnosis of cancer
* Any unstable medical illnesses
* Lifetime history of bipolar disorder, schizophrenia, or psychotic disorder
* Current or recent (past 3 months) substance abuse or dependence
* Current or recent (past 3 months) clinical depression
* Currently taking any medications that have/may have unfavorable interactions with Flibanserin

Ages: 21 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cacioppo, PhD, Principal Investigator — University of Chicago; Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bianchi-Demicheli F, Cojan Y, Waber L, Recordon N, Vuilleumier P, Ortigue S. Neural bases of hypoactive sexual desire disorder in women: an event-related FMRI study. J Sex Med. 2011 Sep;8(9):2546-59. doi: 10.1111/j.1743-6109.2011.02376.x. Epub 2011 Jun 30. PMID 21718449
- [Background] Bolmont M, Cacioppo JT, Cacioppo S. Love is in the gaze: an eye-tracking study of love and sexual desire. Psychol Sci. 2014 Sep;25(9):1748-56. doi: 10.1177/0956797614539706. Epub 2014 Jul 16. PMID 25031302
- [Background] Cacioppo S, Bianchi-Demicheli F, Frum C, Pfaus JG, Lewis JW. The common neural bases between sexual desire and love: a multilevel kernel density fMRI analysis. J Sex Med. 2012 Apr;9(4):1048-54. doi: 10.1111/j.1743-6109.2012.02651.x. Epub 2012 Feb 21. PMID 22353205
- [Background] Cacioppo S, Cacioppo JT. Dynamic spatiotemporal brain analyses using high-performance electrical neuroimaging, Part II: A step-by-step tutorial. J Neurosci Methods. 2015 Dec 30;256:184-97. doi: 10.1016/j.jneumeth.2015.09.004. Epub 2015 Sep 10. PMID 26363189
- [Background] Cacioppo S, Couto B, Bolmont M, Sedeno L, Frum C, Lewis JW, Manes F, Ibanez A, Cacioppo JT. Selective decision-making deficit in love following damage to the anterior insula. Curr Trends Neurol. 2013;7:15-19. PMID 25382944
- [Background] Cacioppo S, Weiss RM, Runesha HB, Cacioppo JT. Dynamic spatiotemporal brain analyses using high performance electrical neuroimaging: theoretical framework and validation. J Neurosci Methods. 2014 Dec 30;238:11-34. doi: 10.1016/j.jneumeth.2014.09.009. Epub 2014 Sep 20. PMID 25244954
- [Background] Ortigue S, Bianchi-Demicheli F. The chronoarchitecture of human sexual desire: a high-density electrical mapping study. Neuroimage. 2008 Nov 1;43(2):337-45. doi: 10.1016/j.neuroimage.2008.07.059. Epub 2008 Aug 13. PMID 18761412

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants started the trial and received the intervention.
Groups:
- Flibanserin: Drug: Flibanserin
  * 8 weeks
  * 100mg once daily at bedtime
  Flibanserin: Observational study using electroencephalogram (EEG) and eye movement tracking device at baseline, week 4, and week 8 while subjects are taking either Flibanserin or matching placebo.
Period: Overall Study
Arm/Group | Flibanserin | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data was collected or analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: EEG Results: Evoked Brain Potentials (Measured Brain Response That is the Direct Result of a Specific Cognitive Event)
Description: Change from baseline EEG results at 8 weeks. Average the electrical brain activity evoked by each type of stimuli to calculate the evoked brain potentials (any stereotyped electrophysical response to a stimulus).
Time Frame: 8 weeks
Population: No data was collected or analyzed
Arm/Group | Flibanserin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Eye Movement Tracking: Movements to First Saccades
Description: Change from baseline eye movement tracking results at 8 weeks.
Time Frame: 8 weeks
Population: No data was collected or analyzed
Arm/Group | Flibanserin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Flibanserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT02770768/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT02770768/ICF_001.pdf